CLINICAL TRIAL: NCT05581264
Title: Effect of Diabetes Self-Management Educational Program on Diabetes Self-Care Activities, Illness Perceptions, Medication Adherence, Health-Related Quality of Life, and Glycemic Control in Patients With Poorly Controlled Type 2 Diabetes
Brief Title: Diabetes Self-Management Educational Program
Acronym: DSMEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mutah University (Other)
Responsible Party: Principal Investigator, Omar Alkhawaldeh, associate professor, Mutah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 120-14-388
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Self-Care Activities; Illness Perceptions; Medication Adherence; Health Related Quality of Life; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Intervention Model Description: This study is a two-arm - experimental vs. control group Randomized Controlled Trial. The sampling frame was patients with uncontrolled type 2 diabetes registered in two outpatient diabetes clinics located in two cities in Jordan. Diabetes self-management program is delivered by a trained diabetes educator facilitator in diabetes management. In addition to the usual care, the intervention group was provided with an education program that consisted of nine 60-min sessions, which included face-to-face interactive sessions with the dissemination and presentation of written and visual materials. The education and counseling were maintained through follow-up (24 weeks) via phone for the intervention group. The control group received only usual care and they were followed according to the institution's diabetes follow-up protocol.
Who Masked: Participant, Outcomes Assessor
Masking Description: To reduce performance bias after the randomization process, blinding is adopted. However, due to the conflicting requirements of ethical and methodological aspects in designing a randomized controlled trial with a psychosocial intervention, double-blinding and randomizing each individual participant posits a huge challenge. Patients and outcome assessors were blinded in a way that none of them will know which group is considered the experimental group and the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Management Education Program (Experimental): Participants received the diabetes self-management education program. The education and counseling were maintained through follow-up via phone for the intervention group
  Interventions: Behavioral: Diabetes Self-Management Education Program
- No Intervention/Control Group (No Intervention): Participants received the usual medical care prescribed by the patient's attending doctor.

INTERVENTIONS:
Behavioral: Diabetes Self-Management Education Program — diabetes self-management education and counseling program with follow-up via phone for the intervention group for 24 weeks
  Arms: Self-Management Education Program

SUMMARY:
Diabetes mellitus is the third most prevalent chronic disease globally. It is a metabolic disorder characterized by elevated blood glucose because of impaired insulin production, reduced insulin effectiveness, or both. It is a major contributor to physical disability and impaired quality of life. Diabetes Self-Management programs help to control blood glucose, reduce hospitalization, and increase compliance; however, the program is underutilized in primary care settings globally, due to cognitive, financial, behavioral, and emotional factors. Addressing the increasing trend in diabetes, Jordan is currently in need of a diabetes self-management program that promotes patient empowerment and overall well-being. The primary aim of this study was to investigate the effectiveness of a diabetes self-management education program for patients with type 2 diabetes in improving self-care, medication adherence, illness perception, health-related quality of life, and glycemic control (HbA1c level). This study is a two-arm randomized controlled trial study of patients with type 2 diabetes attending two outpatients' diabetes clinic settings in Jordan. The education program and also usual medical care were applied to the intervention group, only usual medical care was applied to the control group.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a growing public health problem highly amenable to prevention and health promotion interventions. Diabetes mellitus is a chronic disease that requires ongoing medical care and ongoing patient self-management education and support to prevent acute complications and reduce the risk of chronic complications of diabetes. The prevalence of diabetes mellitus is reaching epidemic proportions in many parts of the world. Globally it is estimated that approximately 537 million adults (20-79 years) are living with diabetes according to International Diabetes Federation (2021). The total number of people living with diabetes is projected to rise to 643 million by 2030 and 783 million by 2045. Moreover, the International Diabetes Federation estimated that diabetes caused at least USD 966 billion dollars in health expenditure - 9% of total spending on adults. In Jordan, the age-standardized prevalence rate of diabetes and impaired fasting blood glucose was 17.1% and 7.8%, respectively. The high prevalence of diabetes point to the need for immediate implementation of educational programs and other interventions to prevent and control the burden of diabetes in Jordan. The majority of researchers and clinicians advocate that diabetes is a disease that requires diabetes self-management care abilities and that patients need to be taught diabetes self-management skills to become reliable, capable, and sufficiently responsible to take care of themselves. Diabetes self-management is of great importance because the adoption of healthy lifestyle behaviors will produce optimum glycemic control for diabetes, which in turn will help minimize or prevent subsequent acute and long-term complications of the disease. Diabetes is a lifelong disease that needs behavioral changes, most often through education, counseling, and support through behavioral interventions offered by health care providers, to enable diabetic patients to perform self-care activities. Behavioral changes are complex processes that are influenced by such factors as illness perceptions, quality of life, beliefs, attitudes, skills, motivation, and social support. In Jordan, diabetes nursing education services are at an early stage of development and have recently been introduced to healthcare facilities and the implementation of such services is still limited. Improving diabetes self-management, preventing diabetes complications, and reducing health service utilization for patients with diabetes are ongoing challenges for nurses and other healthcare providers globally and in Jordan. There is a need to investigate the impact of implementing a nursing educational care program on reaching glycemic control goals and other clinical outcomes because of the increasing prevalence of diabetes and the limited implementation of effective nursing services for patients with type 2 diabetes in Jordan. The primary aim of this study is to evaluate the effect of a structured diabetes education program on glycemic control and other health-related clinical outcomes in patients with poorly controlled type 2 diabetes. This study is a two-arm randomized controlled trial of patients with type 2 diabetes attending two outpatient diabetes clinic settings in Jordan. The education program for 24 weeks and also usual medical care were applied to the intervention group, only usual medical care was applied to the control group.

The education intervention consists of structured face-to-face individual/ group-based education and counseling sessions with telephone follow-up instructions. At each clinic visit, diabetes nurse educators meet the participants in the intervention group in a private room. Printed educational material was developed by the researchers containing information about diabetes, diabetes medications, lifestyle modifications, and self-care activities also given to patients in the intervention group. Diabetes nurse educators also encourage patients to adhere to prescribed medications and advise participants to follow healthy lifestyle behaviors. Finally, follow-up telephone calls were made by the diabetes nurse educator to each intervention participant to discuss and review the prescribed therapy, to emphasize the importance of adherence to the treatment plan, and to answer patient questions or address their concerns. The education and counseling were maintained through follow-up via phone for the intervention group. The control group was not exposed to the structured education intervention but continued with their usual care provided by the medical and nursing staff and was followed according to the institution's routine diabetes follow-up protocol. The baseline assessment (pre-intervention) for both groups involves obtaining data about study outcome measures. The primary outcomes are glycemic control (HbA1c level) and self-care activities; whereas medication adherence, illness perception, and health-related quality of life are the secondary outcomes. Follow-up assessment involves obtaining data about HbA1c results for both the intervention group and the control group from their medical records at 3 and 6 months intervals. The baseline questionnaires were re-administered at six months post-intervention for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years
* Patients with a known diagnosis of type 2 diabetes for at least one year
* Patients with HbA1c >7%, for uncontrolled diabetes
* Able to read, write, and speak Arabic
* Having the ability of autonomous behavior, informed consent, and voluntary participation in the study.
* Receiving oral antidiabetic and/or insulin therapy
* Able to communicate and does not have hearing, speech or psychiatric problems that prevent communication
* Receiving care at one of the participating diabetes clinics

Exclusion Criteria:

* Has an acute or terminal illness or serious mental illness or physical deterioration
* Has any other severe medical conditions that might make it difficult to attend educational sessions
* Planning to travel for longer than 6 weeks during the 6-month intervention period
* Patients not willing to participate in the study
* Type 1 diabetes mellitus, gestational diabetes mellitus, and other special types of diabetes
* Patients who were unable to provide a consent form
* Patients who have hearing, speech, and psychiatric problems that prevent communication
* Cognitive impairment and/or learning disabilities
* Recruited in other research and/or diabetes educational programs during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Difference in diabetes self-care behaviors scale scores between experimental group and control group across time | Baseline, Week 24
  Diabetes Self-Management Questionnaire (DSMQ) DSMQ was used to measure the patient's self-care behaviors. Respondents will be asked to rate their specific self-care activities of last 3 months on a 16-item DSMQ.This questionnaire involves a four point likert scale (ranging from 0 - 'does not apply to me' to 3 - 'applies to me very much'). There are 4 subscales of this study tool; namely, 'Glucose Management' which is comprised of 5 items, 'Dietary Control' comprised of 4 items, 'Physical Activity comprised of 3 items, and, 'Health-Care Use' comprised of 3 items. Higher scores will represent more effective self-care.
Difference in Glycated hemoglobin (HbA1c) level between experimental group and control group across time | baseline, Week 12, Week 24
  HbA1c was analyzed from a sample of venous blood. HbA1c < 7.0% is considered as the good glycemic control and HbA1c ≥ 7.0% will be considered as poorly controlled glucose level

SECONDARY OUTCOMES:
Difference in illness perception scale scores between experimental group and control group across time | Baseline, Week 24
  The Brief Illness Perception Questionnaire (IPQ) was used to measure illness perception. The Brief IPQ has nine items, all of which are rated using a 0-10 response scale except the causal question. Five of the items assess cognitive illness representations: consequences (item 1), with higher scores representing a stronger belief that the illness will have serious consequences; timeline (item 2), with higher scores indicating a belief that the illness is going to last for a longer time; personal control (item 3) and treatment control (item 4), with higher scores indicating a higher level of belief in control or potential for cure of the illness; identity (item 5). Two of the items assess emotional representations: concern (item 6) and emotions (item 8), with higher scores indicating greater worries about health status. One item assesses illness comprehensibility (item 7), with higher scores indicating better understanding of the illness.
Difference in medication adherence scale scores between experimental group and control group across time | Baseline, Week 24
  Self-reported medication adherence (Morisky Scale) was used to measure medication adherence. This scale assessed the probability that patients take their medications as prescribed. The Morisky Scale is an 8-item questionnaire with seven yes/no questions and one question answered on a 5-point Likert scale. Scores range from zero to eight and are categorized into three levels of adherence: 8=high adherence; 6-7=medium adherence; <6=low adherence. The Morisky scale has been used across many chronic diseases, including diabetes, as a self-reported measure of adherence to medications and has demonstrated good reliability and predictive validity.
Difference in health related quality of life HRQOL scale scores between experimental group and control group across time | baseline, Week 24
  The Short-Form 36-item survey (SF-36) was used to assess the HRQOL. The SF-36 is a self-assessment scale, consisting of 36 questions under eight subscales: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Subscale scores are calculated according to standard procedures, yielding score values of 0 to 100, where higher scores indicate better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Omar A Alkhawaldeh, Principal Investigator — Mutah University
Locations (1):
- Diabetes Outpatient Clinic, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The individual participant data has been recorded in an anonymous format digitally and for the sake of confidentiality, participant data will not be shared according to IRB Committee guidelines. However, data will be disseminated in the form of publications, conferences, and presentations. Nevertheless, data may be shared on official request after consultation with the research team and IRB Committee.